CLINICAL TRIAL: NCT00737321
Title: Mechanisms Regulating Wound Vascularization
Status: Terminated | Type: Observational
Why Stopped: investigator moved institutions and did not transfer study
Sponsor: Gayle Gordillo (Other)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0051
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Wounds and Injuries
Keywords: Impact of ischemia; Impact of stress and; Identify patterns of gene expression
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participnts with wounds will have 3 mm punch biopsy performed twice or three times in the whole study period.Obtained tissue sample will be processed immidiately and frozen in liquid nitrogen.The tissue sample will transport to research lab for genomic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2- Diabetics without wound (s): These group of subject will be control arm, included who have good glycemic control diabetic with HbA1c 8.4 or lower and also without any open wounds. Samples will be collected.
  Interventions: Procedure: Samples will be collected
- 1-Subjects with diabetes with wound: This group of subjects will have wound and come for couple of follow up visits for saliva collection, biopsy collection and blood draw.

INTERVENTIONS:
Procedure: Samples will be collected — wound tissue biopsy, blood samples, saliva collection and wound VAC sponge (if applicable).
  Groups: 2- Diabetics without wound (s)

SUMMARY:
This pilot study is designed to assess the impact of ischemia/ diminished wound vascularization and stress on wound healing by comparing patterns of gene expression in specific cell types critical to wound healing biology, e.g. macrophages or endothelial cells.

DETAILED DESCRIPTION:
Chronic wounds affect approximately 2% of the U.S. population at any given time. Animal models can not simulate the complex set of pre-existing conditions in each individual that results in failed wound healing. Therefore, human subjects must be used to obtain valid data. Adequate wound vascularization that permits blood vessels to deliver oxygen to the wound is a requirement for wound healing to occur. This protocol will attempt to gain greater understanding of the mechanisms of chronic wounds through 3 specific aims: 1) identify the angiogenic mechanisms in wound site macrophages, which are required for healing, 2) determine the impact of stress and glucocorticoid resistance on endothelial cell and macrophage biology and ultimately wound healing outcomes, 3) identify patterns of gene expression in wound endothelial cells that are found in healing versus non-healing wounds. This data will be correlated with the wound oxygenation status to determine the impact of wound vascularization on the observed biological responses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years
* ischemic wound group
* non-ischemic wound group
* diabetes with good glycemic control
* lower extremity wound

Exclusion Criteria:

* Age greater ≥ 70 years
* End stage renal disease
* Unable to provide informed consent
* Pregnant women
* Therapeutically anticoagulated
* Prisoners
* Periwound TcOM < 25mmHg
* Spinal cord injury
* Taking immunosuppressive medications
* Individuals with current diagnosis of a major psychiatric illness (e.g.schizophrenia,psychosis)
* Severe protein malnutrition- pre-albumin < 10 mg/dl or albumin < 2 g/dl
* Diabetes with poor glucose control-defined as hgb A1c > 8.4%

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (n=80)including controlled group will be recruited from the OSU outpatient wound care center located at Morehouse plaza and OSU East, OSU plastic surgery, OSU diabetic clinics.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in Gene Expression Profile in Healing versus Non-healing Wounds | 12 weeks
  Wound tissue biopsies, saliva, serum samples and wound sponges will be obtained at an initial time point, at the midpoint of the study and near the end of wound closure over a 12 week window. If the wound closes quickly, i.e. less than 4 weeks then only 2 biopsies will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - OSU East Wound Care Center, Columbus, Ohio
  - OSU Comprehensive Wound Care Center Morehouse, Columbus, Ohio

REFERENCES:
- [Result] Beckrich K, Aronovitch SA. Hospital-acquired pressure ulcers: a comparison of costs in medical vs. surgical patients. Nurs Econ. 1999 Sep-Oct;17(5):263-71. No abstract available. PMID 10711175